CLINICAL TRIAL: NCT06174844
Title: Evaluation and Development of the HUMANisation of CARE in the Andalusian Public Health System in Complex User Units and Hospital Emergency Units: Attention to Frailty, Prevention of Adverse Events, and the Impact of the Nurse-patient Relationship on Health Outcomes
Brief Title: Assessment of the Humanisation of Care in Hospitals in Andalusia-Spain
Acronym: HUMANCUIDA
Status: Recruiting | Type: Observational
Sponsor: University of Seville (Other)
Collaborators: Andalusian Health Service (Other Government)
Responsible Party: Principal Investigator, REGINA ALLANDE CUSSO, Principal Investigator, University of Seville
Other Study IDs: PI22/00373
Record Dates: First submitted 2023-12-06; First posted 2023-12-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: PROM; Satisfaction, Patient; Satisfaction, Personal; Stress; Burnout, Professional; Hospital Acquired Condition; Adverse Event; Nurse-Patient Relations
Keywords: Humanization of care; Health outcomes
MeSH Terms: conditions — Patient Satisfaction; Personal Satisfaction; Burnout, Professional; Iatrogenic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sample 1: Data collected from 1st January to 30th June of 2024
  Interventions: Other: No intervention applied
- Sample 2: Data collected from 1st January to 30th June of 2025
  Interventions: Other: No intervention applied

INTERVENTIONS:
Other: No intervention applied — No intervention applied: data will only be collected in the indicated sampling periods from patients admitted to the participating hospitals.

SUMMARY:
Observational assessment through patient interviews of relational, structural and organisational aspects related to the humanisation of health care. These data will be related to health outcomes such as pain, sleep quality, anxiety levels, adverse events (pressure injuries, falls, and mortality), satisfaction with the care received, and experience in communication processes with health professionals.

Data will also be collected on work ergonomics variables (stress, burnout, working conditions, ratios) of nurses and health technicians, which will also be related to the health outcomes collected.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the internal medicine and emergency units of the participating hospitals during the sampling time.

Exclusion Criteria:

* Patients presenting with haemodynamic instability or emergencies at the time of sampling
* Patients with cognitive impairment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the internal medicine and emergency units of the participating hospitals during the sampling time
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Health outcomes | 12 months
  Levels obtained in the health outcomes identified as study variables: anxiety, measured with the Golberg scale; sleep quality, measured with the Athens Sleep Scale; frailty status, measured with the Tilburg Index; level of pain, measured with the Visual Analogue Pain Scale; level of care dependency, measured with the INICIARE scale; and the variables of mortality, falls, venous catheter infection and pressure injuries, which will be asked with items created ad-hoc. We will also study the association between the results obtained with the aforementioned scales and the variables of organisational context and structure of the centre: management leadership, measured with the Leadership Scale; nurse-patient relationship, measured with the NIC_CA Scale; work stress, measured with the Nursing Stress Scale; work conditions, measured with the PES-NWI Scale; and the variables of turnover intention and nurse-patient ratio, measured with questions designed ad hoc.
Adverse events | 12 months
  Design of a predictive model based on regression models of the occurrence of adverse events (falls, mortality, venous catheter infection pressure injuries, which will be asked with items created ad-hoc) and their relationship with the rest of the study variables (assessed with the scales used for outcome 1).

CONTACTS AND LOCATIONS:
Overall Officials: Regina Allande-Cussó, Dr., Principal Investigator — Andalusian Health Service and University of Seville
Locations (1):
- Hospital Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
The collected data is personal and will not be shared or publicized. These data will be stored by the research team for 10 years, following the specifications of the Ethics Committee that approved the Ethical opinion.

REFERENCES:
- [Derived] Allande-Cusso R, Mejias-Martin YA, Quinoz-Gallardo MD, Porcel-Galvez AM. The impact of humanising hospital care on health outcomes: an observational study protocol. BMC Nurs. 2025 Apr 28;24(1):463. doi: 10.1186/s12912-025-03105-w. PMID 40296139